CLINICAL TRIAL: NCT05945498
Title: Randomized, Double-blind, Placebo-controlled Phase 1 Trial of ТВ/Flu-05Е Intranasal Vector Vaccine for the Prevention of Tuberculosis Infection in BCG-vaccinated Volunteers Aged 18-50
Brief Title: Evaluation of ТВ/Flu-05Е Vaccine for the Prevention of Tuberculosis Infection in BCG-vaccinated Volunteers Aged 18-50 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tatyana Zubkova (Other)
Responsible Party: Sponsor-Investigator, Tatyana Zubkova, Head of the clinical department, Research Institute of Influenza, Russia
Organization: Research Institute of Influenza, Russia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ВПТ-II-01/2022
Record Dates: First submitted 2023-06-13; First posted 2023-07-14 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Tuberculosis Infection
Keywords: Tuberculosis infection; Vaccine; BCG boost; Influenza vector
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TB/Flu-05E vaccine (Experimental): Single dose of 7.7 lg EID50 vector vaccine
  Interventions: Biological: TB/Flu-05E vaccine
- Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TB/Flu-05E vaccine — Participants will receive single intranasal injection of A/H1N1pdm09 recombinant attenuated influenza vector (7.7 lg EID50) with modified NS gene coding for the TB10.4 and HspX antigens of M. tuberculosis
  Arms: TB/Flu-05E vaccine
Biological: Placebo — Participants will receive single intranasal injection of placebo buffer solution
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate safety, reactogenicity and immunogenicity of the TB/Flu-05E single-dose intranasal vaccine for the prevention of Tuberculosis infection in BCG-vaccinated Volunteers aged 18-50 years.

DETAILED DESCRIPTION:
Study include 51 participants in two cohorts. At the first stage, 15 volunteers (Cohort 1), randomized in a 2:1 ratio (10 people in the vaccine group and 5 people in the placebo group) will be included in the study. At the second stage, the following 36 people (Cohort 2) will be included in the study, which will be randomly distributed (randomization) in a ratio of 2: 1 for the vaccine preparation (24 people) and placebo (12 people). Duration of the study for each participant is about 4 months (no more than 122 days).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy BCG-vaccinated men and women aged 18 to 50 years
2. Availability of signed informed consent
3. Diagnosed "healthy" according to the data of standard clinical, laboratory and instrumental examination methods, with the absence of clinically significant changes. Participants with chronic conditions that do not require special treatment, such as diabetes mellitus, hypertension, or heart disease, are eligible to participate in this study if the investigator considers the participant's condition to be medically stable
4. The ability and willingness to make entries in the diary of self-observation, as well as to carry out all the visits foreseen in the study for control medical observation
5. Consent to use effective contraceptive methods throughout their participation in the study.
6. Body weight ≥ 50 kg
7. HI antibody titers ≤1:20 to influenza A/H1N1pdm09
8. Negative test for alcohol in exhaled air
9. Consent to use effective contraceptive methods throughout their participation in the study
10. Values of the complete blood count and biochemical blood analysis (during the screening) within 0.9*reference range lower limit and 1,1 * reference range upper limit
11. Negative tests for HIV, hepatitis B, hepatitis C, and syphilis

Exclusion Criteria:

1. Participation in another clinical study within three months prior to the start of the current study; planning to participate in another study during the current study period
2. Clinical, radiological or laboratory signs of active or previously transferred tuberculosis of any localization.
3. Passage in the past or at the present time of examination in anti-tuberculosis medical institutions
4. Existence in the past or present of contact with patients with any form of tuberculosis (at home, at work, in the circle of friends and acquaintances)
5. Tuberculous infection confirmed by the TB-FERON IGRA laboratory test
6. Immunization with BCG within six months prior to enrollment in the current study
7. Contact with COVID-19 patients within 14 days prior to the start of the clinical study
8. Positive rapid test result for SARS-CoV-2 antigen
9. Immunization with any other non-study vaccine product within three weeks prior to enrollment in the current study, or refusal to postpone such until the end of the three-week period after completion of the current study
10. Regular use of nasal irrigation therapy during the last six months prior to enrollment in the current study or episodic use of the above method of treatment in the two weeks prior to the screening
11. History of frequent nosebleeds (>5) during the year prior to the current study
12. Clinically significant anatomic pathology or the presence of surgical intervention in the sinus area, paranasal sinuses, or traumatic injuries of the nose within a month before screening
13. Symptoms of acute respiratory disease, including fever, or other acute illness at the time of screening or within two weeks prior to screening
14. Treatment with immunoglobulins or other blood derived medications in the three months prior to screening or planning such treatment during the period of participation in the current study; donation of blood/plasma (450 ml or more) less than 2 months prior to screening
15. The presence or suspicion of the presence of various immunosuppressive or immunodeficiency conditions or continuous use (the drug was prescribed for more than 14 days without a break) of immunosuppressive drugs, immunomodulators for 6 months before the screening (for corticosteroids, ≥0.5 mg/kg per day of prednisone or other corticosteroid equivalent; topical and inhaled steroids).
16. History of bronchial asthma
17. Hypersensitivity and the presence of severe allergic reactions, including Quincke's edema, anaphylactic shock after the previous administration of any vaccine
18. History of wheezing after previous immunization with live influenza vaccine
19. Other adverse events after immunization (fever above 40°C, syncope, non-febrile convulsions, anaphylaxis) when there is a minimal likelihood that they are associated with a previous administration of any vaccine
20. Suspicion of hypersensitivity to any component of the study vaccine, including egg protein
21. Seasonal (in spring or autumn) increased sensitivity to the effects of natural factors
22. Acute or chronic clinically significant lung, cardiovascular, hepatic, endocrine, neurological, or psychiatric disorders, or impaired renal function identified by history, physical examination, or clinical laboratory findings that, in the opinion of the investigator, may influence the outcome of the study
23. History of leukemia or any other malignant diseases of the blood or solid malignant neoplasms of other organs
24. History of thrombocytopenic purpura or bleeding disorders
25. History of convulsions
26. The presence or suspicion of the presence of various immunosuppressive or immunodeficiency conditions, including HIV infection
27. Tuberculosis or residual changes after tuberculosis according to the anamnesis and / or available medical documentation
28. Chronic alcohol dependence or chronic use of illicit drugs, drug abuse
29. Claustrophobia and social phobia according to history and / or available medical records
30. For women of reproductive age - lactation, pregnancy or suspected pregnancy, early postpartum period
31. Premenopausal women (last menstrual period <1 year prior to signing informed consent) who are not surgically sterile and women who are of reproductive potential but do not use or plan to use valid birth control throughout the study and do not agree to perform a urine pregnancy test while participating in the study
32. Military personnel undergoing military service on conscription
33. Persons in custody in pre-trial detention centers and serving sentences in places of deprivation of liberty
34. Special diet (eg, vegetarian, vegan, salt-restricted) or lifestyle (night work, extreme physical activity)
35. Any condition that, in the opinion of the investigator, may increase the risk to the health of a volunteer participating in the study or affect the results of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with local and systemic adverse events (AEs) and serious adverse events (SAEs) | Throughout the study, average of 4 months
  Number of participants with AEs and SAEs including those of particular interest:
  * immediate AEs (allergic reactions) occurring within 2 h after vaccination;
  * post-vaccination reactions between 2 h and a subsequent 7 days;
  * other AEs including unexpected clinical manifestations of a local and systemic nature occurring on the day of vaccination and the following 7 days;
  * influenza A virus shedding detected by rapid test in nasal swab samples

SECONDARY OUTCOMES:
Concentration of cytokines in nasal secrets after vaccination | Days 1, 2, 3
  Change from baseline in the concentration of cytokines in nasal secrets measured in ELISA (pg/ml, 13-plex assay, IFN-α2, TSLP, IL-1α, IL-1β, GM-CSF, IL-11, IL-12p40, IL-12p70, IL-15, IL-18, IL-23, IL-27, IL-33)
Level of mucosal IgA antibody in nasal secret/saliva | Days 1, 21
  Titers of IgA antibody measured in ELISA in nasal secret/saliva
Level of TB antigen-specific cytokine producing T-cells | Days 1, 7, 21
  Change from baseline in the level of cytokine producing T-cells upon in vitro stimulation of PBMC with M. tuberculosis peptide epitopes measured by ICS/ELISPOT
Level of influenza specific cytokine producing T-cells | Days 1, 7, 21
  Change from baseline in the level of cytokine producing T-cells upon in vitro stimulation of PBMC with А/H1N1pdm09 influenza measured by ICS/ELISPOT
Level of TB antigen-specific cytokine release in whole blood assay | Days 1, 7, 21
  Change from baseline in the cytokine concentration in whole-blood cytokine release assay upon in vitro stimulation with M. tuberculosis peptide epitopes measured in ELISA
Level of А/H1N1pdm09 influenza specific cytokine release in whole blood assay | Days 1, 7, 21
  Change from baseline in the cytokine concentration in whole-blood cytokine release assay upon in vitro stimulation with А/H1N1pdm09 influenza measured in ELISA
Level of TB antigen-specific IgG antibody | Days 1, 21
  Changes in the levels of TB antigen-specific total serum IgG antibodies measured in ELISA in serum
Influenza specific local antibody immune response | Days 1, 21
  Change from baseline in the level of influenza specific IgA antibodies in nasal secret/saliva measured in ELISA
Influenza specific systemic antibody immune response | Days 1, 21
  Change from baseline in the titer of influenza specific antibodies in serum measured in hemagglutination inhibition/microneutralisation assay

CONTACTS AND LOCATIONS:
Locations (1):
- Smorodintsev Research Institute of Influenza, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No